CLINICAL TRIAL: NCT02236572
Title: A Neoadjuvant Phase II Trial of Aromatase Inhibitors in Combination With Everolimus in Postmenopausal Women With Hormone Receptor Positive/HER2 Negative Breast Cancers With Low and Intermediate Risk (< 25) Oncotype Dx Recurrence Scores
Brief Title: Neoadj ph 2 AI Plus Everolimus in Postmenopausal Women w/ ER Pos/HER2 Neg, Low Risk Score
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Phase 2 of recruitment was contingent on 5 of 15 patients responding, which did not occur.
Sponsor: Yale University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1405013982
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Results first posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer
Keywords: Postmenopausal; ER-positive, PR-positive, HER2-negative; Low and intermediate risk
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aromatase Inhibitor plus Everolimus (Experimental): Aromatase inhibitor plus everolimus by mouth daily for 26 weeks
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Aromatase inhibitor plus everolimus by mouth daily for 26 weeks. All patients will begin treatment on Cycle 1 Day 1 with both the standard dose of one of the following 3 aromatase inhibitors ( physician's choice) plus everolimus 10 mg by mouth daily:
  * Anastrozole 1 mg
  * Letrozole 2.5 mg
  * Exemestane 25 mg

SUMMARY:
The purpose of this study is to see whether adding everolimus to hormone treatment before breast surgery will increase the chances of shrinking the breast cancer in those patients with hormone-responsive breast cancer and a lower Oncotype DX® Recurrence Score ( 25 or less), compared to prior experience with hormone therapy alone. Everolimus is a drug currently approved for use by the United States Food and Drug administration (FDA) for the treatment of patients with advanced or metastatic kidney or breast cancer. Everolimus is considered investigational for non-metastatic breast cancer patients.

DETAILED DESCRIPTION:
This is a single arm open-labeled neoadjuvant phase II clinical trial evaluating everolimus in combination with an aromatase inhibitor in postmenopausal women with hormone receptor positive/HER2 negative breast cancers with low and intermediate risk (< 25) Recurrence Scores by Oncotype Dx.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of hormone receptor positive, HER2 negative invasive breast carcinoma.
* Tumors must be estrogen and/or progesterone receptor positive according to ASCO/CAP 2010 guidelines as either ER or PR ≥ 1% positive nuclear staining by immunohistochemistry. Estrogen and/or progesterone receptor results by Oncotype Dx will not be accepted.
* Tumors must be HER2 negative as defined according to ASCO/CAP 2013, as HER2 0 - 1+ by IHC or non-amplified FISH or CISH. If HER2 IHC is 2+, FISH/CISH must be performed and must not be positive (must be a ratio of < 2), but otherwise FISH/CISH is not required if IHC is 0 or 1+ by institutional standards.
* Patients must not have had prior ipsilateral breast-conserving surgery or total mastectomy and be eligible for neoadjuvant treatment.
* Clinical Stage II-IIIC (T2-4 N0-3 M0) by mammogram, ultrasound or MRI
* Baseline Oncotpye Dx recurrence score < 25.
* Staging studies with a CT scan of the chest and abdomen and bone scan, or a PET/CT is required for clinical stage III, and are considered optional for stage II breast cancers.
* Patients with multifocal, multicentric and synchronous bilateral breast cancers are allowed:

  * Multifocal disease is defined as more than one invasive cancer < 2 cm from the largest lesion within the same breast quadrant.
  * Multicentric disease is defined as more than one invasive cancer ≥ 2 cm from the largest lesion within the same breast quadrant or more than one lesion in different quadrants.
  * Synchronous bilateral disease is defined as invasive breast cancer in both breasts, diagnosed within 30 days of each other.
  * In patients with multicentric or bilateral invasive breast cancers, all sampled lesions must be hormone receptor-positive and HER2-negative. Any lesion measuring > 1 cm must have an Oncotype Dx and the score must be < 25. Lesions less than 1 cm in size are not required to have an Oncotype Dx. One lesion (typically the largest) should be designated as the target lesion for which clinical and radiographic response to the neoadjuvant therapy will be judged.
  * Patients with a hormone receptor-positive, HER2-negative invasive cancer that meets study criteria may have ductal carcinoma in situ in another quadrant of the same breast or in the contralateral breast even if the DCIS is hormone receptor-negative.
* Patients must have adequate bone marrow function, as defined by peripheral granulocyte count of ≥ 1,500/mL, hemoglobin ≥ 9 g/dL and a platelet count ≥ 100,000/ mL within 28 days prior to registration.
* Patients must have adequate hepatic function obtained within 28 days prior to registration and documented by all of the following:

  * Bilirubin ≤ 1.5 mg/dL (or ≤ 3.0 mg/dL if due to Gilbert's Syndrome)
  * ALT and AST ≤ 1.5 x Institutional Upper Limit of Normal (IULN)
  * Alkaline phosphatase ≤ 1.5 x IULN
* Patients must have adequate renal function with serum creatinine level ≤ IULN within 28 days prior to registration.
* Patients must have a fasting cholesterol ≤ 300 mg/dl OR ≤7.75 mmol/L and triglycerides ≤ 2.5 x IULN obtained within 28 days prior to registration. Patients may be on lipid lowering agents to reach these values.
* Patients must have a ECOG performance status of 0-2.
* Patients must be able to take oral medications.
* Postmenopausal women (women are considered post-menopausal and not of child-bearing potential if they are > 18 years of age and have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms or biochemically postmenopausal by estradiol and FSH levels) prior to enrollment, or have had surgical bilateral oophorectomy (with or without hysterectomy) prior to registration. Medical ovarian suppression with LHRH agonists to render a patient postmenopausal will not be acceptable.

  16. Patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent prior to any screening procedures in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Patients must not have inflammatory breast cancer (T4d) and must not have metastatic breast cancer (Stage IV disease).
* Patients must not have prior exposure to mTOR inhibitors (e.g. rapamycin, everolimus, sirolimus, temsirolimus, deforolimus).
* Patients must not have prior treatment with any investigational drug within the preceding 28 days and must not be planning to receive any other investigational drug for the duration of the study.
* Patient may not have any impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of the drug (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).
* Uncontrolled diabetes mellitus as defined by HbA1c >8% within 28 days prior to registration despite adequate therapy.
* Patients who have any severe and/or uncontrolled cardiac disease within ≤ 6 months prior to start of everolimus, including: unstable angina pectoris, Symptomatic congestive heart failure of New York heart Association Class III or IV, myocardial infarction, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease
* Patients must not have an organ allograft or other history of immune compromise.
* Patients must not be receiving chronic, systemic treatment with corticosteroids or other immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* Patients must not have a known history of HIV seropositivity
* Patients must not have a known diagnosis of hepatitis B or C. Patients with the following risk factors must have hepatitis screening pre-treatment:

  * Blood transfusions prior to 1990
  * Current or prior IV drug users
  * Current or prior dialysis
  * Household contact with a hepatitis B or C patient
  * Current or prior high-risk sexual activity
  * History of jaundice.
* Patients must not have any known uncontrolled underlying pulmonary disease or severely impaired lung function (spirometry and DLCO 50% or less of normal and O2 saturation 88% or less at rest on room air),
* Active (acute or chronic) or uncontrolled severe infection.
* Patients who have received live attenuated vaccines within 1 week of start of Everolimus, or have plans to receive such vaccination while on protocol treatment. Patient should also avoid close contact with others who have received live attenuated vaccines. Examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines;
* Patients who are currently part of or have participated in any clinical investigation with an investigational drug within 1 month prior to dosing;
* Patients must not have taken within 14 days prior to registration , be taking, nor plan to take while on protocol treatment, strong CYP3A4 inhibitors, and/or CYP3A4 inducers.
* Patients with active bleeding diathesis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-11-29 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lajos Pusztai, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Aromatase Inhibitor Plus Everolimus: Aromatase inhibitor plus everolimus by mouth daily for 26 weeks
  Everolimus: Aromatase inhibitor plus everolimus by mouth daily for 26 weeks. All patients will begin treatment on Cycle 1 Day 1 with both the standard dose of one of the following 3 aromatase inhibitors ( physician's choice) plus everolimus 10 mg by mouth daily:
  * Anastrozole 1 mg
  * Letrozole 2.5 mg
  * Exemestane 25 mg
Period: Overall Study
Arm/Group | Aromatase Inhibitor Plus Everolimus
Started | 17
Completed | 14
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Aromatase Inhibitor Plus Everolimus
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 66 [54 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10
  Black | 3
  Multiple or unknown | 4
Region of Enrollment [Number; unit: participants]
  United States | 17
Clinical Tumor Size at Presentation - pt no. [Count of Participants; unit: Participants] — Clinical size was defined as the largest diameter on contrast-enhanced computed tomography. The higher the number (e.g. T1 compared to T3), the greater the progression.
  Participants
    T1 | 5
    T2 | 12
    T3 | 0
Nodal Status at Presentation [Count of Participants; unit: Participants] — Nodal Status at Presentation: Lymph node status shows whether or not the lymph nodes in the underarm area (axillary lymph nodes) contain cancer:
  * Lymph node-negative means none of the axillary lymph nodes contain cancer.
  * Lymph node-positive means at least one axillary lymph node contains cancer.
  Participants
    Positive (biopsy proven) | 2
    Negative | 15
Tumor Histology [Count of Participants; unit: Participants] — A description of a tumor based on how abnormal the cancer cells and tissue look. Examples include; Ductal carcinoma in situ (DCIS), Lobular carcinoma in situ, Invasive ductal carcinoma (ductal breast cancer)
  Participants
    Ductal | 12
    Lobular | 3
    Unknown | 2

OUTCOME MEASURES:

1. Primary Outcome: Achievement of a PEPI Score of 0 Following Neoadjuvant Treatment With Everolimus and an Aromatase Inhibitor
Description: (PEPI) preoperative endocrine prognostic index. The total PEPI score assigned to each patient is the sum of the risk points derived from the pT stage, pN stage, Ki67 level, and estrogen receptor status of the surgical specimen. An HR in the range of 1-2 receives one risk point; a HR in the 2-2.5 range, two risk points; a HR greater than 2.5, three risk points. The total risk point score for each patient is the sum of all the risk points accumulated from the four factors in the model. A lower PEPI score indicates lower risk for recurrence. A score of 0 is lowest risk for recurrence.
Time Frame: up to 26 weeks
Population: 15 patients had surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Aromatase Inhibitor Plus Everolimus
Number analyzed (Participants) | 15
Participants
  PEPI Score = 0 | 4
  PEPI Score > 0 | 11

2. Secondary Outcome: PEPI Score
Description: To obtain the PEPI score, risk points for relapse-free survival (RFS) are assigned depending on the hazard ratio (HR) from the multivariable analysis. The total PEPI score assigned to each patient is the sum of the risk points derived from the pT stage, pN stage, Ki67 level, and estrogen receptor status of the surgical specimen. A HR in the range of 1 to 2 receives one risk point; a HR in the 2 to 2.5 range, two risk points; a HR greater than 2.5, three risk points. The total risk point score for each patient is the sum of all the risk points accumulated from the four factors in the model, ranges from 0 (best possible outcome) to 12 (worst possible outcome).
Time Frame: up to 26 weeks
Population: Those that completed surgery
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Aromatase Inhibitor Plus Everolimus
Number analyzed (Participants) | 15
units on a scale | 3 [0 to 7]

3. Secondary Outcome: Participant Ability to Tolerate Study Treatment With Minimal Side Effects
Description: Adverse events (using CTCAE (4.0)) that begin or worsen after informed consent were recorded. Adverse events are itemized in the adverse events module (in terms of total events and total participants experiencing events). Presented are the total number of participants that experience adverse events. For clarification, counts of participants that experienced serious adverse events and counts of participants that experienced 'other' (not serious) adverse events are presented separately.
Time Frame: Up to 26 weeks
Population: All participants that were enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Aromatase Inhibitor Plus Everolimus
Number analyzed (Participants) | 17
Participants
  Participants with Serious Adverse Events | 5
  Participants with Other (Not Including Serious) Adverse Events | 17

ADVERSE EVENTS:
Time Frame: Up to 26 weeks
Arm/Group | Aromatase Inhibitor Plus Everolimus
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 5/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aromatase Inhibitor Plus Everolimus (N=17)
Atrial Flutter (Cardiac disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aromatase Inhibitor Plus Everolimus (N=17)
Fatigue (General disorders) | 10 (16)
Edema limbs (General disorders) | 7 (8)
Pain (General disorders) | 6 (9)
Edema face (General disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2)
General disorders and administration site conditions - Other (General disorders) | 1 (2)
Malaise (General disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 12 (22)
Nausea (Gastrointestinal disorders) | 6 (7)
Diarrhea (Gastrointestinal disorders) | 5 (9)
Constipation (Gastrointestinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 7 (10)
Cholesterol high (Investigations) | 7 (11)
Alanine aminotransferase increased (Investigations) | 6 (8)
Platelet count decreased (Investigations) | 3 (4)
Weight loss (Investigations) | 3 (5)
Investigations - Other (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1)
INR increased (Investigations) | 1 (5)
Neutrophil count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (20)
Anorexia (Metabolism and nutrition disorders) | 5 (10)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 5 (5)
Hypokalemia (Metabolism and nutrition disorders) | 5 (6)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 (13)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 7 (7)
Headache (Nervous system disorders) | 6 (6)
Dizziness (Nervous system disorders) | 4 (4)
Paresthesia (Nervous system disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (9)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 9 (13)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Vascular disorders) | 5 (26)
Hot flashes (Vascular disorders) | 4 (5)
Urinary tract infection (Infections and infestations) | 2 (2)
Bronchial infection (Infections and infestations) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Blurred vision (Injury, poisoning and procedural complications) | 1 (1)
Eye disorders - Other (Injury, poisoning and procedural complications) | 1 (1)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-16): https://cdn.clinicaltrials.gov/large-docs/72/NCT02236572/Prot_SAP_000.pdf